CLINICAL TRIAL: NCT06918340
Title: Evaluation of Analgesic Efficacy of Lidocaine and Diclofenac Spray in Radial Artery Blood Gas Sampling by Visual Analogue Scale (VAS) and Perfusion Index: A Randomised, Placebo-Controlled Study
Brief Title: Evaluation of Analgesic Efficacy of Lidocaine and Diclofenac Spray in Radial Artery Blood Gas Sampling by Visual Analogue Scale and Perfusion Index
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sinem Dogruyol, Associate Professor Doctor, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-KAEK-64
Record Dates: First submitted 2025-03-28; First posted 2025-04-09 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Blood Gas Analysis; Topical Analgesia
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Topical treatments will be administered in 100 cc amber coloured glass spray bottles to ensure blinding in all three treatment groups. The bottles will be prepared by the responsible investigator and numbered with the number on the sealed envelope. Thus, it will be ensured that the treating staff and the patient will be blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I: 5-6 puffs of topical 10% lidocaine spray (Active Comparator): Group I: 5-6 puffs of topical 10% lidocaine spray will be applied before radial artery blood gas sampling.
  Interventions: Drug: Lidocaine spray
- Group II: topical 1% diclofenac spray (Active Comparator): Group II: 5-6 puffs of topical 1% diclofenac spray will be applied before radial artery blood gas sampling.
  Interventions: Drug: Diclofenac
- Group III: topical 70% alcohol solution spray (Placebo Comparator): Group III: 5-6 puffs of topical 70% alcohol solution spray will be applied before radial artery blood gas sampling.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Diclofenac — Group II: 5-6 puffs of topical 1% diclofenac spray will be applied before radial artery blood gas sampling.
  Arms: Group II: topical 1% diclofenac spray
Drug: Lidocaine spray — Group I: 5-6 puffs of topical 10% lidocaine spray will be applied before radial artery blood gas sampling.
  Arms: Group I: 5-6 puffs of topical 10% lidocaine spray
Other: Placebo — Group III: 5-6 puffs of topical 70% alcohol solution spray will be applied before radial artery blood gas sampling.
  Arms: Group III: topical 70% alcohol solution spray

SUMMARY:
The aim of this clinical trial is to evaluate the analgesic efficacy of lidocaine and diclofenac sprays to be administered before the procedure in cases admitted to the emergency department and requiring radial artery blood gas sampling by means of visual pain scale (VAS) and perfusion index in comparison with placebo. The main questions it aims to answer are:

1. Is there a difference between the efficacy of two different sprays? 2. Is there a significant difference between the side effects of two different sprays? Researchers will compare diclofenac sodium, lidocain and placebo sprays. Treatments will;

1. be administered in same three spray bottles to ensure blinding in the groups.
2. Randomisation will be done by closed envelope method.
3. Numerical Pain Scale (NRS) will be used to evaluate the analgesic efficacy of the sprays. NRS scores will be recorded in both groups before starting blood gas sampling (baseline) and after blood gas sampling.
4. Any side effects due to medication will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65.
* Having clinical indication for radial artery blood gas sampling
* Being conscious, co-operative and orientated
* Those who approved the informed consent form

Exclusion Criteria:

* Being under 18 years of age.
* Being pregnant or breastfeeding.
* Not being conscious, co-operative and orientated (impaired consciousness)
* Being used painkillers in the last 24 hours
* Radial artery blood gas sampling on the same day (more than one application)
* Presence of cardiac arrhythmia
* Have a diagnosis of neuropathy (including diabetic neuropathy)
* Having a diagnosis of anxiety and panic disorder
* Using a sustained-release dermal analgesic patch (fentanyl)
* Patient unable to comply with the visual analogue pain scale (VAS) due to language barrier
* Presence of a condition such as dementia, etc. that may lead to a change in consciousness
* Allergy to lidocaine or diclofenac

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores associated with radial artery blood gas sampling | Baseline perfusion index and baseline VAS will be measured and recorded. 10 minutes after blood gas sampling, perfusion index and VAS score will be recorded.
  The primary outcome of the study was the change in pain associated with radial artery blood gas sampling. It is aimed to provide patient comfort with spray applications. Differences between the 3 groups in VAS scores related to the intervention will be analysed.

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpasa Numune Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: SAP, ICF, CSR
Time Frame: 12 months ( 01.01.2025-01.01.2026)
Access Criteria: The researcher responsible for data analysis will be authorised to access IPD for 1 year.

REFERENCES:
- [Derived] Altundag I, Dogruyol S, Yavuz BG, Afacan MA, Colak S. 10% Lidocaine Versus 1% Diclofenac Spray in Radial Arterial Blood Gas Sampling: A Randomized, Double-Blind, Placebo-Controlled Trial using Perfusion Index. J Emerg Med. 2025 Dec 16;81:39-47. doi: 10.1016/j.jemermed.2025.12.015. Online ahead of print. PMID 41576782